CLINICAL TRIAL: NCT06113627
Title: Prevention-Related Lymphatic Response to Resistance Exercise in Breast Cancer Survivors at Risk of Breast Cancer-Related Lymphedema
Brief Title: Lymphatic Response to Resistance Exercise in Breast Cancer Survivors
Acronym: LinfoGYM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Cristina Roldán-Jiménez, Profesor and Reseacher (PT, PhD), University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-2023
Record Dates: First submitted 2023-10-09; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer Lymphedema; Survivorship; Lymphedema of Upper Limb
Keywords: Breast Cancer; Lymphedema, Early-Onset; Breast Cancer Lymphedema; Exercise Therapy; Exercise Training; Acute Exercise; Exercise Movement Techniques; Physiotherapy (Techniques)
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of the researchers in charge of the evaluations and data analysis will be implemented, so that they are unaware of the assignment of each patient to the groups. It is not possible to blind participants and the physiotherapist (care provider) due to the very nature of the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The intervention group will receive a total of 24 sessions of Therapeutic Resistance Exercise, distributed in 2 weekly sessions of 50 minutes during 3 months.
  Interventions: Other: Resistance Therapeutic Exercise
- Control group (No Intervention): The control group will receive an educational booklet containing generalized mobility exercises such as frontal and lateral shoulder raises and rotations (hands to head, hands behind back). This is usually the usual treatment, since in most centers, patients are only referred for treatment of LACM when it is already established.

INTERVENTIONS:
Other: Resistance Therapeutic Exercise — Strength exercises will be aimed at large muscle groups, such as the shoulder, chest, back and also muscle groups of the lower extremities. In the initial 2 weeks, intervention will start with low intensities of around 55-65% of 1RM, which allows to perform around 15-20 repetitions. The first week there will be performed 2 series, while in the second week it will be 3 series.
  Moderate intensity in the 2nd week, corresponding to 65-75% of 1RM and allowing for around 8-12 repetitions. 3 series will be maintained throughout this period of time.In addition to the progressive change in intensity, throughout the intervention the load will be increased by 5-10% when the patient performs the exercise too easily or when they can perform more repetitions than estimated. Rest between sets will be 2-3 minutes.
  Arms: Exercise group

SUMMARY:
The objective of this study is 1) to study the acute and chronic effect of resistance therapeutic physical exercise (RTPE) in the prevention of breast cancer-related lymphedema (BCRL) in breast cancer survivors at risk using variables related to the lymphatic response; 2) Study the possible relationship between changes in body composition at a local and regional level and volume changes produced by RTPE in patients at risk of suffering from BCRL.

DETAILED DESCRIPTION:
Nowadays, research studies that confirm the safety and preventive effect of resistance or strength exercise in breast cancer-related lymphedema (BCRL) have been limited to the study of changes in variables related to the lymphatic response, such as bioimpedance spectroscopy , X-ray absorptiometry, perometry or water displacement after completion of a resistance exercise program (chronic effect).

To better understand the preventive effect of resistance exercise on the BCRL, in addition to studying the variables that are globally accepted and studied at a regional level such as the volume due to water displacement, variables that measure changes at a regional level related to body composition, such as such as echogenicity and ultrasound thickness, local tissue water and mechanical properties of tissues. Furthermore, this would allow us to detect possible changes in different body regions of the upper quadrant (upper extremity, but also breast or back), and not only taking global changes into account. On the other hand, the lymphatic response should be studied in the short term (acute effect), in the long term after an exercise program (chronic effect), as well as in the short term after the training period with possible adaptations to the lymphatic system that could explain the preventive effect.

Therefore, although there is a strong degree of scientific evidence to include therapeutic strength physical exercise as a preventive tool for LACM, the possible physiological mechanisms involved are unknown. The aim of the present project is to tudy the acute and chronic effect of resistance therapeutic physical exercise (RTPE) in the prevention of breast cancer-related lymphedema (BCRL) in breast cancer survivors at risk using regional but also local variables related to the lymphatic response, as well as to study between changes in these variables, body composition at a local and regional level and volume changes produced by RTPE in breast cancer survivors at risk of suffering from BCRL

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer
* Being of legal age
* Histologically confirmed primary Breast Cancer (I-IIIA) (without the presence of metastasis) with a diagnosis in the last year
* Unilateral involvement
* Surgery for the tumor at least 6 weeks before the start of the intervention
* WHO performance status of 0 (asymptomatic, complete and ambulatory activity)
* Correct understanding of Spanish
* Approval by signing the informed consent;
* Mus be considered at risk for developing LACM: 1) Have undergone surgery that includes axillary dissection; 2) Have received or are undergoing regional lymph node radiation; 3) BMI >30 kg/m2. . These patients are considered to have stage 0, subclinical or latent according to the International Society of Lymphology (ISL) , since they will not present signs or symptoms, but lymphatic transport will be altered by the treatments themselves

Exclusion Criteria:

* Women already diagnosed with LACM in stage I, II or III according to the ISL or if they present an L-Dex ratio > 10 or a difference in volume equal to or greater than 10% between both extremities
* Suffer from or have been diagnosed with any other lymphatic-venous disease in the upper extremity, such as venous insufficiency, thrombosis or lipedema;
* Suffer from conditions that prevent resistance exercise of the upper body
* Participation in regular (>1 time/week) and intense exercises involving the upper extremity during the last month
* Suffer from heart disease
* Inability to complete questionnaires;
* A physical condition that prevents them from making hospital visits
* Taking any drug that may affect the lymphatic and circulatory system, such as diuretics or corticosteroids
* Women which presents some type of wound or infection on the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Changes in volume difference between extremities (%) | Six measures: Baseline, before and 24 hours after the day 5 of exercise session, before and 24 hours after the 24 day of exercise session; after 3 month once completed the whole intervention, and after 1 year
  The volume of both extremities will be measured to obtain the difference between both, which will be used as a relative criterion to determine the preventive effect of the intervention, determining the appearance of LACM as those cases in which the patient reaches a difference after one year of follow-up. volume equal to or greater than 10% between both extremities. It will be measured using water displacement volumetry, considered the gold standard for measuring the volume of the affected limb.

SECONDARY OUTCOMES:
Changes in extracelular fluid (ECF) | Six measures: Baseline, before and 24 hours after the day 5 of exercise session, before and 24 hours after the 24 day of exercise session; after 3 month once completed the whole intervention, and after 1 year
  The EFC of the affected and contralateral side (liters, l) will be obtained. Which will allow establishing the ECF radius between the extremities. This ratios will be allowed to estimate L-Dex. The L-Dex ratio ranges between -10 and +10, taking into account the ratio between the dominant and non-dominant arms, which is equivalent to impedance ratios of 0.935 to 1.139 for the dominant arms at risk and from 0.862 to 1.066 for non-dominant arms at risk, respectively. It will be obtained through bioimpedance spectroscopy
Changes in Percentage Water Content (PWC) | Six measures: Baseline, before and 24 hours after the day 5 of exercise session, before and 24 hours after the 24 day of exercise session; after 3 month once completed the whole intervention, and after 1 year
  Local tissue water will be measured by bilateral tissue dielectric constant (TDC). values on the forearm and biceps using the MoistureMeterD Compact. PWC%= 100%x(TDC-1)/77.5. It will be measured on the anterior and posterior aspects of the arm and forearm, on the breast, on the lateral aspect of the shoulder and in the dorsal area.
Changes in Thickness of the dermis and subdermis | Six measures: Baseline, before and 24 hours after the day 5 of exercise session, before and 24 hours after the 24 day of exercise session; after 3 month once completed the whole intervention, and after 1 year
  It will be obtained through the analysis of ultrasound images. The thickness will be measured in millimeters (mm). It will be measured on the anterior and posterior aspects of the arm and forearm, on the breast, on the lateral aspect of the shoulder and in the dorsal area.
Changes in echogenicity of the dermis and subdermis | Six measures: Baseline, before and 24 hours after the day 5 of exercise session, before and 24 hours after the 24 day of exercise session; after 3 month once completed the whole intervention, and after 1 year
  It will be obtained through the analysis of ultrasound images. Echogenicity or echointensity refers to the average value obtained from a histogram generated from an 8-bit gray scale. This analysis does not have units of measurement, but provides a numerical value between 0 and 255. It will be measured on the anterior and posterior aspects of the arm and forearm, on the breast, on the lateral aspect of the shoulder and in the dorsal area.
Changes in elastic properties of tissues. | Six measures: Baseline, before and 24 hours after the day 5 of exercise session, before and 24 hours after the 24 day of exercise session; after 3 month once completed the whole intervention, and after 1 year
  It will be measured with a MyotonPRO portable device (Myoton AS, Estonia), whose probe will be placed on the surface of the skin and produce a mechanical stimulus that will provide five parameters: Tone (Hz), Dynamic stiffness (N/m), Elasticity (unit relative), Relaxation time (ms) and Fluency (relative unit). It will be measured on the anterior and posterior aspects of the arm and forearm, on the breast, on the lateral aspect of the shoulder and in the dorsal area.
Quality of life (QoL) | Six measures: Baseline, before and 24 hours after the day 5 of exercise session, before and 24 hours after the 24 day of exercise session; after 3 month once completed the whole intervention, and after 1 year
  it will be measured using the European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life questionnaire (EORTC QLQ-BR23). This is an EORTC QLQ-C30 breast cancer module that contains 23 items that assess disease symptoms, treatment side effects, body image, sexual functioning, and future outlook. All items are rated on a 4-point scale (1, not at all to very much). Higher scores represent better functioning and higher symptom scores show greater problems. Cronbach's α ranged from 0.46 to 0.94, showing high reliability.
Active Range of Movement (AROM, degrees) | Six measures: Baseline, before and 24 hours after the day 5 of exercise session, before and 24 hours after the 24 day of exercise session; after 3 month once completed the whole intervention, and after 1 year
  Abduction and flexion of the shoulder joint complex will be measured. It will be measured in a sitting position, ensuring that there is no movement of the trunk, using a digital inclinometer.
Grip strength (kg) | Three measures: Baseline , after 3 month once completed the whole intervention (post-intervention) and after 1 year (follow-up)
  It will be measured using the Jamar Hydraulic Hand dynamometer. All participants will sit in a chair without armrests, with their feet on the floor and their back straight, holding the dynamometer with their dominant arm. The elbow was flexed at 90° and the wrist was in a neutral position (0°). Maximum isometric voluntary contractions will be performed for 5 seconds. The force will be expressed in kg. Of the 3 measurements carried out, the peak force will be recorded in units of Newtons (N) or in Kilograms (Kg), obtained from both extremities
Perceived shoulder function (%) | Three measures: Baseline , after 3 month once completed the whole intervention (post-intervention) and after 1 year (follow-up)
  It will be measured using the Shoulder Pain and Disability Index (SPADI) questionnaire. SPADI consists of 13 items that are distributed in two different subscales: one related to pain, which contains 5 items, and another related to disability, which contains 8 items. Scoring of items in both subscales is on a scale ranging from 0 (indicating absence of pain or disability) to 10 (representing the worst pain imaginable or such significant difficulty in performing tasks that help is needed). The higher the score on each subscale, the greater the pain intensity and the greater the disability experienced by the individual evaluated.
Symptoms Related to Lymphedema | Three measures: Baseline , after 3 month once completed the whole intervention (post-intervention) and after 1 year (follow-up)
  It will be measured using the Spanish version of the Breast Cancer and Lymphedema Symptom Experience Index (BCLE-SEI) questionnaire.This questionnaire consists of 2 parts: Part 1 is made up of 24 items and evaluates the symptoms of LACM using a Likert scale from 0 (absence of a certain symptom) to 4 (greater severity of a certain symptom); Part 2 is made up of 32 items that evaluate the symptom of discomfort, that is, the negative impact and suffering evoked by the experience of lymphedema. Each part is calculated with the sum of all the responses, and in turn they can be added together to obtain a total score
Fear-Avoidance | Three measures: Baseline , after 3 month once completed the whole intervention (post-intervention) and after 1 year (follow-up)
  It will be measured using the Spanish version of Fear-Avoidance component scale (FACS). The FACS contains 20 separate items that are scored from 0 ("completely disagree") to 5 ("completely agree"), with a total possible score of 100. Five severity levels are available for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80), and ex- treme (81-100). This questionnaire has been validated in breast cancer population, showing good psychometric properties.

CONTACTS AND LOCATIONS:
Locations (1):
- Cristina Roldán Jiménez, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roldán-Jiménez C. What are the physiologic effects of Resistance Exercise behind breast cancer-related lymphedema prevention? Medical Hypotheses Volume 171, February 2023, 111022. https://doi.org/10.1016/j.mehy.2023.111022
- [Background] Roldan-Jimenez C, Pajares B, Ruiz-Medina S, Trinidad-Fernandez M, Gonzalez-Sanchez M, Ribelles N, Garcia-Almeida JM, Rios-Lopez MJ, Alba E, Cuesta-Vargas AI. Design and implementation of a standard care programme of therapeutic exercise and education for breast cancer survivors. Support Care Cancer. 2022 Feb;30(2):1243-1251. doi: 10.1007/s00520-021-06470-9. Epub 2021 Aug 31. PMID 34463835
- [Background] Gutierrez-Sanchez D, Pajares-Hachero BI, Trinidad-Fernandez M, Escriche-Escuder A, Iglesias-Campos M, Bermejo-Perez MJ, Alba-Conejo E, Roldan-Jimenez C, Cuesta-Vargas A. The Benefits of a Therapeutic Exercise and Educational Intervention Program on Central Sensitization Symptoms and Pain-Related Fear Avoidance in Breast Cancer Survivors. Pain Manag Nurs. 2022 Aug;23(4):467-472. doi: 10.1016/j.pmn.2022.01.003. Epub 2022 Mar 9. PMID 35277360
- [Background] Roldan-Jimenez C, Martin-Martin J, Pajares B, Ribelles N, Alba E, Cuesta-Vargas AI. Factors associated with upper limb function in breast cancer survivors. PM R. 2023 Feb;15(2):151-156. doi: 10.1002/pmrj.12731. Epub 2021 Nov 23. PMID 34713595
- [Background] Escriche-Escuder A, Trinidad-Fernandez M, Pajares B, Iglesias-Campos M, Alba E, Cuesta-Vargas AI, Roldan-Jimenez C. Ultrasound use in metastatic breast cancer to measure body composition changes following an exercise intervention. Sci Rep. 2021 Apr 23;11(1):8858. doi: 10.1038/s41598-021-88375-5. PMID 33893370
- [Background] Davies C, Levenhagen K, Ryans K, Perdomo M, Gilchrist L. Interventions for Breast Cancer-Related Lymphedema: Clinical Practice Guideline From the Academy of Oncologic Physical Therapy of APTA. Phys Ther. 2020 Jul 19;100(7):1163-1179. doi: 10.1093/ptj/pzaa087. PMID 32589208
- [Background] Wang L, Shi YX, Wang TT, Chen KX, Shang SM. Breast cancer-related lymphoedema and resistance exercise: An evidence-based review of guidelines, consensus statements and systematic reviews. J Clin Nurs. 2023 May;32(9-10):2208-2227. doi: 10.1111/jocn.16437. Epub 2022 Jul 27. PMID 35894167